CLINICAL TRIAL: NCT06663527
Title: Compound Phellodendron Decoction May Promote Wound Healing After Anal Fistulotomy
Acronym: CPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Heng Deng, The Second Affiliated Hospital of Anhui University of Chinese Medicine, The Second Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-zj-19; 2023AH050848 (Other Grant/Funding Number: cientific Research Project of Colleges and Universities of Anhui Province)
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2024-10

CONDITIONS: Fistula in Ano
Keywords: Anal fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): Study group (n=30) treated fumigating-washing therapy with the CPD
  Interventions: Combination Product: Fumigating-washing Therapy With CPD
- Control Group (Placebo Comparator): Control group (n=30) underwent fumigating-washing therapy with a placebo
  Interventions: Combination Product: fumigating-washing therapy with a placebo

INTERVENTIONS:
Combination Product: Fumigating-washing Therapy With CPD — All patients underwent anal fistulectomy based on the Parks classification. For postoperative infection prophylaxis, cefuroxime was used at a dosage of 2g per dose, twice daily. Commencing the day following surgery, a fumigating-washing therapy was conducted once daily either after defecation or two hours prior to intravenous infusion. In the study group, a medical solution used for fumigating-washing therapy was prepared by blending 200 ml of CPD with 2 liters of water at 40 °C. This medicinal solution was then transferred into the reservoir of an ultrasonic atomizing fumigating-washing device (Model:TM50-C, Xuzhou Tianma Medical Equipment Factory, China) that was classified by the FDA as Class II (special controls).
  Arms: Study Group
Combination Product: fumigating-washing therapy with a placebo — fumigating-washing therapy with a placebo
  Arms: Control Group

SUMMARY:
Sitz-bath therapy with Chinese medicine has significant advantages in the management of postoperative wounds of anal fistula. This method not only ensures safety, efficacy, and cost-effectiveness, but also simplifies application. With a firm foundation in a historical heritage, this method is notable for their minimal adverse reactions. The fumigating-washing or sitz-bath therapy with Compound Phellodendron Decoction (CPD) for postoperative wounds of anal fistula has demonstrated efficacy in mitigating pain, reducing edema, curbing secretions, alleviating skin itching, and promoting wound healing processes. Despite the body of clinical research in this domain is substantial, the majority of studies have been limited to observing therapeutic outcomes. The intrinsic mechanisms by which these effects are achieved remain elusive. This study aims to unravel the potential mechanisms underpinning CPD's promotion of wound healing, focusing on the aspects of inflammation and immunity.

ELIGIBILITY:
Inclusion Criteria:age range of 18 to 80 years who had undergone anal fistulotomy procedures.

-

Exclusion Criteria:patients with Crohn's disease, pregnancy or lactation, organ dysfunction (such as heart failure, respiratory insufficiency, liver or renal impairment, gastrointestinal dysfunction), coagulopathy, autoimmune diseases, or a history of hypersensitivity to Chinese medicinal substances.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-26 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
The healing duration of wounds | The healing duration of wounds, edema, exudation, and pain scores, served as the principal observation index.
  The healing duration of wounds, edema, exudation, and pain scores, served as the principal observation index.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui university of Chinese Medicine, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided